CLINICAL TRIAL: NCT05315713
Title: A Phase Ib/II Open-Label, Multicenter Study Evaluating the Safety, Efficacy, and Pharmacokinetics of Mosunetuzumab in Combination With Tiragolumab With or Without Atezolizumab in Patients With Relapsed or Refractory B-Cell Non-Hodgkin Lymphoma
Brief Title: An Open-Label, Multicenter Study Evaluating the Safety, Efficacy, and Pharmacokinetics of Mosunetuzumab in Combination With Tiragolumab With or Without Atezolizumab in Participants With B-Cell Non-Hodgkin Lymphoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to Sponsor decision.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO43116
Record Dates: First submitted 2022-03-31; First posted 2022-04-07 (Actual); Results first posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-09

CONDITIONS: Non-Hodgkin Lymphoma, Follicular Lymphoma
Keywords: B-Cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Follicular; Lymphoma, B-Cell | interventions — Tiragolumab; atezolizumab; tocilizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Subcutaneous (SC) Mosunetuzumab in Combination with Intravenous (IV) Tiragolumab (Experimental): Participants will receive at least 8 and up to 17 cycles of treatment (cycle length = 21 days)
  Interventions: Drug: Mosunetuzumab SC; Drug: Tiragolumab; Other: Tocilizumab
- Mosunetuzumab SC in Combination with Tiragolumab IV and Atezolizumab IV (Experimental): Participants will receive at least 8 and up to 17 cycles of treatment (cycle length = 21 days)
  Note: This arm did not enroll any participants.
  Interventions: Drug: Mosunetuzumab SC; Drug: Tiragolumab; Drug: Atezolizumab; Other: Tocilizumab

INTERVENTIONS:
Drug: Mosunetuzumab SC — Participants will receive SC mosunetuzumab for up to 17 treatment cycles (cycle length = 21 days)
Drug: Tiragolumab — Participants will receive IV tiragolumab every 3 weeks (Q3W) for up to 17 treatment cycles (cycle length = 21 days)
Drug: Atezolizumab — Participants will receive IV atezolizumab Q3W for up to 17 treatment cycles (cycle length = 21 days)
  Arms: Mosunetuzumab SC in Combination with Tiragolumab IV and Atezolizumab IV
Other: Tocilizumab — Participants will receive IV tocilizumab as needed to manage cytokine release syndrome (CRS) events

SUMMARY:
This study will evaluate the safety, efficacy, and pharmacokinetics of mosunetuzumab in combination with tiragolumab, with or without atezolizumab, in participants with relapsed or refractory (R/R) diffuse large B-cell lymphoma (DLBCL) or follicular lymphoma (FL) who have received at least two previous lines of systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Aged >/= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Life expectancy of at least 12 weeks
* Histologically documented FL or DLBCL that has relapsed or failed to respond to at least two prior systemic treatment regimens and for which no suitable therapy of curative intent or higher priority exists (e.g., standard chemotherapy, ASCT, CAR T cells)
* At least one bi-dimensionally measurable (> 1.5 cm) nodal lesion, or at least one bi-dimensionally measurable (> 1.0 cm) extranodal lesion
* Participants with FL (including trFL) for whom a bone marrow biopsy and aspirate can be collected
* Adequate hematologic and organ function

Exclusion Criteria:

* Received any of the following treatments prior to study entry: mosunetuzumab or other CD20/CD3-directed bispecific antibodies; tiragolumab or other anti-TIGIT agent; allogenic SCT; solid organ transplantation
* Currently eligible for autologous SCT
* Current or past history of CNS lymphoma or leptomeningeal infiltration
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibody therapy (or recombinant antibody-related fusion proteins)
* Contraindication to atezolizumab (if applicable) or tocilizumab
* Clinically significant toxicities from prior treatment have not resolved to Grade </= 1 (per NCI CTCAE v5.0) prior to the first study drug administration with exceptions defined by the protocol
* Treatment-emergent immune-mediated adverse events associated with prior immunotherapeutic agents as defined by the protocol
* Evidence of any significant, concomitant disease as defined by the protocol
* Major surgery within 4 weeks prior to first study treatment administration, with the exception of protocol-mandated procedures (e.g., tumor biopsies and bone marrow biopsies)
* Significant cardiac, pulmonary, CNS, or liver disease, or known active infections
* History of other malignancy that could affect compliance with the protocol or interpretation of results
* History of autoimmune disease with exceptions as defined in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2023-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (17):
- United States (3):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - University of Michigan, Ann Arbor, Michigan
  - Lifespan Cancer Institute, Providence, Rhode Island
- Australia (3):
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Eastern Health, Box Hill, Victoria
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
- Belgium (4):
  - AZ Sint Jan Brugge Oostende AV, Bruges
  - Institut Jules Bordet, Brussels
  - AZ Groeninge, Kortrijk
  - CHU UCL Namur - Mont-Godinne, Yvoir
- Canada (2):
  - Tom Baker Cancer Centre-Calgary, Calgary, Alberta
  - Princess Margaret Cancer Centre, Toronto, Ontario
- Universitaet Duisburg-Essen, Essen, Germany
- United Kingdom (4):
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Royal Marsden Hospital - Institute of Cancer Research - Chelsea, London
  - Plymouth Hospitals NHS Trust - Derriford Hospital, Plymouth
  - Royal Marsden Hospital - Institute of Cancer Research - Sutton, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Groups:
- Subcutaneous (SC) Mosunetuzumab in Combination With Intravenous (IV) Tiragolumab: Participants received SC mosunetuzumab on Cycle (C) 1 Day (D) 1, C1D8, C1D15, and on the first day of each subsequent 21-day treatment cycle. Participants also received IV tiragolumab every 3 weeks (Q3W).
Period: Overall Study
Arm/Group | Subcutaneous (SC) Mosunetuzumab in Combination With Intravenous (IV) Tiragolumab
Started | 8
Completed | 0
Not Completed | 8
Not completed — Death | 5
Not completed — Progressive disease | 1
Not completed — Withdrawal by Subject | 1
Not completed — Study terminated by sponsor | 1

BASELINE CHARACTERISTICS:
Arm/Group | Subcutaneous (SC) Mosunetuzumab in Combination With Intravenous (IV) Tiragolumab
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.9 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events - Phase 1b
Time Frame: From the start of treatment until 90 days after the final dose of study treatment (up to 36 weeks)
Measure: Number; unit: Percentage of participants
Arm/Group | Subcutaneous (SC) Mosunetuzumab in Combination With Intravenous (IV) Tiragolumab
Number analyzed (Participants) | 8
Percentage of participants | 100

2. Primary Outcome: Best Objective Response Rate (ORR) as Determined by the Investigator Using Lugano 2014 Criteria - Phase 2
Time Frame: Up to Cycle 17 (cycle length = 21 days)
Population: This endpoint was not evaluated due to early study termination (Phase 2 did not occur and no data was collected).
Arm/Group | Subcutaneous (SC) Mosunetuzumab in Combination With Intravenous (IV) Tiragolumab
Number analyzed (Participants) | 0

3. Secondary Outcome: Best ORR as Determined by the Investigator Using Lugano 2014 Criteria - Phase 1b
Description: Best ORR is defined as the fraction of participants with complete response (CR) or partial response (PR) at any time as determined by the investigator using Lugano 2014 criteria.
Time Frame: Assessed at screening and then every 3-6 months until disease progression, start of new anti-cancer therapy, or withdrawal (through Cycle 8; cycle length = 21 days)
Measure: Number; unit: Percentage of participants
Arm/Group | Subcutaneous (SC) Mosunetuzumab in Combination With Intravenous (IV) Tiragolumab
Number analyzed (Participants) | 8
Percentage of participants | 62.5

4. Secondary Outcome: Serum Concentration of Mosunetuzumab - Phase 1b
Time Frame: Cycle 1 Day 1 - Cycle 8 Day 1 (cycle length = 21 days)
Population: The PK population included all participants with at least one serum sample post-dose for mosunetuzumab.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Subcutaneous (SC) Mosunetuzumab in Combination With Intravenous (IV) Tiragolumab
Number analyzed (Participants) | 8
ug/mL
  C1D1 pre-dose | NA (NA) — Pre-dose serum concentrations were below the limit of quantification.
  C1D1 3 hrs post-dose | 0.00983 (NA) — There were insufficient data points above the limit of quantification to calculate the CV.
  C1D2 24 hrs post-dose | 0.0556 (109.6)
  C1D4 72 hrs post-dose | 0.164 (90.5)
  C1D8 pre-dose | 0.166 (83.2)
  C1D15 pre-dose: number analyzed (Participants) | 7
  C1D15 pre-dose | 2.18 (48.8)
  C2D1 pre-dose: number analyzed (Participants) | 7
  C2D1 pre-dose | 4.02 (86.3)
  C3D1 pre-dose: number analyzed (Participants) | 6
  C3D1 pre-dose | 2.90 (81.8)
  C4D1 pre-dose: number analyzed (Participants) | 5
  C4D1 pre-dose | 2.34 (49.0)
  C4D1 3 hrs post-dose: number analyzed (Participants) | 6
  C4D1 3 hrs post-dose | 2.10 (48.2)
  C5D1 pre-dose: number analyzed (Participants) | 4
  C5D1 pre-dose | 2.59 (25.7)
  C8D1 pre-dose: number analyzed (Participants) | 3
  C8D1 pre-dose | 2.97 (17.7)

5. Secondary Outcome: Best Complete Response (CR) Rate as Determined by the Investigator Using Lugano 2014 Criteria - Phase 1b
Time Frame: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Subcutaneous (SC) Mosunetuzumab in Combination With Intravenous (IV) Tiragolumab
Number analyzed (Participants) | 8
Percentage of participants | 37.5

6. Secondary Outcome: Duration of Response (DOR) as Determined by the Investigator Using Lugano 2014 Criteria - Phase 1b and Phase 2
Time Frame: From the first occurrence of a documented response (CR or partial response (PR)) to disease progression or relapse, or death from any cause, whichever occurs first (up to approximately 4 years)
Population: Phase 1b is reported. No data was collected for Phase 2.
Measure: Number; unit: Time
Arm/Group | Subcutaneous (SC) Mosunetuzumab in Combination With Intravenous (IV) Tiragolumab
Number analyzed (Participants) | 5
Time | NA — The endpoint could not be analyzed due to an insufficient number of participants with the event.

7. Secondary Outcome: Progression-Free Survival (PFS) as Determined by the Investigator Using Lugano 2014 Criteria - Phase 2
Time Frame: From the first study treatment to the first occurrence of disease progression or relapse, or death from any cause, whichever occurs first (up to approximately 4 years)
Population: This endpoint was not evaluated due to early study termination (Phase 2 did not occur and no data was collected).
Arm/Group | Subcutaneous (SC) Mosunetuzumab in Combination With Intravenous (IV) Tiragolumab
Number analyzed (Participants) | 0

8. Secondary Outcome: Event-Free Survival (EFS) as Determined by the Investigator Using Lugano 2014 Criteria - Phase 2
Time Frame: as for outcome 7
Population: This endpoint was not evaluated due to early study termination (Phase 2 did not occur and no data was collected).
Arm/Group | Subcutaneous (SC) Mosunetuzumab in Combination With Intravenous (IV) Tiragolumab
Number analyzed (Participants) | 0

9. Secondary Outcome: Overall Survival (OS) - Phase 2
Time Frame: From the time of first study treatment to death from any cause (up to approximately 4 years)
Population: This endpoint was not evaluated due to early study termination (Phase 2 did not occur and no data was collected).
Arm/Group | Subcutaneous (SC) Mosunetuzumab in Combination With Intravenous (IV) Tiragolumab
Number analyzed (Participants) | 0

10. Secondary Outcome: Percentage of Participants With Adverse Events - Phase 2
Time Frame: From the start of treatment until 90 days after the final dose of study treatment
Population: This endpoint was not evaluated due to early study termination (Phase 2 did not occur and no data was collected).
Arm/Group | Subcutaneous (SC) Mosunetuzumab in Combination With Intravenous (IV) Tiragolumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From the start of treatment until 90 days after the final dose of study treatment (up to 36 weeks)
Arm/Group | Subcutaneous (SC) Mosunetuzumab in Combination With Intravenous (IV) Tiragolumab
All-Cause Mortality (participants affected / at risk) | 5/8
Serious Adverse Events (participants affected / at risk) | 2/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subcutaneous (SC) Mosunetuzumab in Combination With Intravenous (IV) Tiragolumab (N=8)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
Pneumonia aspiration (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Cerebellar haematoma (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subcutaneous (SC) Mosunetuzumab in Combination With Intravenous (IV) Tiragolumab (N=8)
Anaemia (Blood and lymphatic system disorders) | 3 (4)
Neutropenia (Blood and lymphatic system disorders) | 2 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Ear congestion (Ear and labyrinth disorders) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Malignant dysphagia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Oral pain (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 2 (2)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Injection site reaction (General disorders) | 3 (4)
Malaise (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 2 (2)
Pyrexia (General disorders) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
Cytomegalovirus infection reactivation (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Rhinovirus infection (Infections and infestations) | 1 (1)
Fractured sacrum (Injury, poisoning and procedural complications) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2)

LIMITATIONS AND CAVEATS:
Early termination led to small numbers of participants for analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-20): https://cdn.clinicaltrials.gov/large-docs/13/NCT05315713/Prot_SAP_001.pdf